CLINICAL TRIAL: NCT01599000
Title: Artemether-Lumefantrine Clinical Effectiveness Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Papua New Guinea Institute of Medical Research (Other Government)
Collaborators: Australian Agency for International Development (Unknown); National Department of Health, Papua New Guinea (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MRAC.09.13
Record Dates: First submitted 2012-04-01; First posted 2012-05-15 (Estimated); Last update posted 2012-08-16 (Estimated); Status verified 2012-08

CONDITIONS: Parasitologically Confirmed; Malarial
Keywords: malaria; Plasmodium; Papua New Guinea; artemether/lumefantrine
MeSH Terms: conditions — Malaria | interventions — Artemether, Lumefantrine Drug Combination; lactitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Efficacy arm (Active Comparator): Supervised administration of six doses of fixed-dose artemether-lumefantrine (Coartem, Novartis)
  Interventions: Drug: Artemether-lumefantrine combination
- Effectiveness arm (Experimental): Un-supervised administration of six doses of fixed-dose artemether-lumefantrine (Coartem, Novartis)
  Interventions: Drug: Artemether-lumefantrine combination

INTERVENTIONS:
Drug: Artemether-lumefantrine combination — fixed-dose tablet, six doses over three days, according to weight group
  Other Names: Coartem, Novartis

SUMMARY:
In 2009, Papua New Guinea officially adopted artemether-lumefantrine (AL) as new national first-line drug for uncomplicated malaria. The principal purpose of this study is to measure the absolute effectiveness of AL when used under real-life clinical conditions, as compared to optimized in-vivo trial conditions. This question was raised by the National Department of Health in preparation for the country-wide roll-out of AL.

The study is designed as a randomized controlled trial comparing two study arms. Patients in the "effectiveness arm" receive the first dose of AL under full supervision in the clinic; the following doses will be taken at home, as in real-life clinical practice and according to the new national treatment guidelines. Patients in the "efficacy arm" will receive all doses of AL as directly observed treatment in the clinic in order to establish the efficacy of the drug when used under ideal conditions.

The study will enroll outpatients aged 6 months to 10 years with a history of fever and a positive rapid test for malaria. Patients meeting all enrollment criteria and providing full written informed consent by a parent/caretaker will be randomized into either of the two study arms. Patients in both arms will be followed up actively for 42 days. Patients in the efficacy arm will be scheduled for visits on days 0, 1, 2, 3, 7, 14, 28 and 42; patients in the effectiveness arm on days 0, 3, 7, 14, 28 and 42.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 months to 10 years (+/- 1 month for children without known date of birth)
* Permanent resident in the study area
* Not enrolled in another study at the same time
* No known history of hypersensitivity reactions to artemether or lumefantrine
* History of fever in the previous 72 hours (approximate)
* Rapid diagnostic test (RDT) positive for any species of Plasmodium

Exclusion Criteria:

* General danger signs: inability to drink or breastfeed, vomiting everything, recent history of convulsions, lethargy or unconsciousness, inability to sit or stand up
* Signs of severe malaria (impaired consciousness, respiratory distress, circulatory collapse, abnormal bleeding, jaundice, or as determined by clinician)
* Severe malnutrition: defined as a child whose weight-for-height is below -3 standard deviation or less than 70% of the median of the NCHS/WHO normalized reference values, or who has symmetrical oedema involving at least the feet; or middle upper arm circumference under 12 cm
* Clinically significant concomitant disease requiring admission
* Contraindications mentioned in the national treatment guidelines

Ages: 6 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 159 (Actual)
Dates: Start 2011-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Adequate Clinical and Parasitological Response (ACPR) | 42 days
  ACPR = Absence of parasitemia on Day 42 irrespective of axillary temperature without previously meeting any of the criteria of Early Treatment Failure or Late Clinical Failure or Late Parasitological Failure (adapted from WHO 2003).

CONTACTS AND LOCATIONS:
Overall Officials: Manuel W Hetzel, PhD, Principal Investigator — Papua New Guinea Institute of Medical Research; Mueller Ivo, PhD, Principal Investigator — Walter and Eliza Hall Institute of Medical Research; Peter M Siba, PhD, Principal Investigator — Papua New Guinea Institute of Medical Research
Locations (1):
- Gurney Health Centre, Alotau, Milne Bay Province, Papua New Guinea